CLINICAL TRIAL: NCT01801839
Title: Detection Of Monocytes/Macrophages Function And Tim-3 Expression In Septic Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jia Li, Medical doctor of Department of Respirtory Disease, Chinese PLA General Hospital
Other Study IDs: 2009BAI86B03
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Sepsis; SIRS(Systemic Inflammatory Response Syndrome)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- SIRS,sepsis,normal: SIRS
  (1) temperature > 38 centigrade or < 36 centigrade; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000/μL or < 4000/μL , or > 10% immature cells.
  sepsis
  SIRS + infection.
  normal
  not SIRS and have no infection.

SUMMARY:
The imbalance between anti- and pro-inflammation often occurs in patients with sepsis. And continuous such imbalance could lead to immunoparalysis, which is characterized by loss of delayed type hypersensitivity, failure of primary infections eradication, and a predisposition of secondary nosocomial infections development. However, in which phase of sepsis does immunoparalysis occur is still unknown. So this study aims to tentatively understand this problem by checking monocytes/macrophages' antigen presentation and cytokine secretion，and by checking monocytes/macrophages' expression of Tim-3 (the T cell transmembrane, immunoglobulin, and mucin-3), which is an inhibitory regulatory molecule, in sepsis patients' peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old;
* Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 ℃ or lower than 36 ℃ (b)respiratory rate above 20/min, or carbon dioxide partial pressure below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.
* Clinically suspected infection;

Exclusion Criteria:

* were under 18 years of age;
* were refused by the patients or his/her familiality;
* were suffering from acquired immunodeficiency syndrome,viral hepatitis,autoimmune diseases and hematology;
* use medicine which can affect immune system,such as Glucocorticoid and Immunosuppressant
* died within 24h after being taken into the ICU, or refused to get involved in the study, or gave up treatment during the period of observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between August 2012 and March 2013 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
systemic inflammatory response to infection with organ dysfunction, hypoperfusion, or hypotension | within 24 hours after enter experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, MD, Study Director — Respiratory Disease Department of Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China